CLINICAL TRIAL: NCT01143142
Title: Vax Facts HPV: Study of a Computer-based Tailoring System and Mothers' Intentions to Vaccinate Their Daughters Against HPV
Brief Title: Vax Facts Human Papillomavirus (HPV): Study of a Computer-based Tailoring System and Mothers' Intentions to Vaccinate Their Daughters Against HPV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Amanda Dempsey, Associate Professor of Pediatrics, University of Colorado, Denver
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 149891; P50CA101451 (NIH)
Record Dates: First submitted 2010-06-10; First posted 2010-06-14 (Estimated); Results first posted 2014-12-22 (Estimated); Last update posted 2014-12-22 (Estimated); Status verified 2014-12

CONDITIONS: Human Papillomavirus; Prevention
Keywords: Human papillomavirus; HPV; Prevention; Tailoring; Persuasive communication; Adolescent

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tailoring (Experimental): Individuals assigned to the experimental group will receive a two-page brochure tailored based on their responses to the survey.
  Interventions: Behavioral: Computer-based tailoring system
- Untailored information (Active Comparator): Individuals assigned to the control group will receive the CDC vaccine information sheet that is standardly provided.
  Interventions: Behavioral: Computer-based tailoring system

INTERVENTIONS:
Behavioral: Computer-based tailoring system — Both the intervention and control groups will use a computer-based tailoring system to respond to survey questions. The computer-based tailoring system will produce messages for a two-page educational brochure based on participants' responses to survey questions. Only the intervention group will receive this brochure.

SUMMARY:
The goal of this study is to determine whether a two-page print brochure that delivers individually tailored educational messages about the Human papillomavirus (HPV) vaccine increases HPV vaccine-hesitant mothers' intentions to have their adolescent daughters vaccinated against HPV.

DETAILED DESCRIPTION:
This will be a randomized controlled intervention trial for HPV vaccine-hesitant mothers of adolescent (ages 11-15 years old) girls. Mothers will complete a three-item measure that assesses their baseline intentions for having their adolescent daughter vaccinated against HPV. Mothers will then fill out a short, computer-based survey that assesses demographic factors, prior experience with HPV-associated illnesses and views about a variety of potential barriers to HPV vaccination. Following the survey, the intervention group (40 mothers) will receive a two-page print brochure that uses their survey data to generate the brochure such that it addresses each mother's top three concerns about the HPV vaccine. The control group (40 mothers) will receive a generic, two-page brochure that is similar in appearance to the intervention, but contains only untailored, generic information about the vaccine. HPV vaccination intention will be assessed a second time after reading the brochure, using the same three-item measure as before the survey. The vaccine administration records of the adolescent daughters of these mothers will be accessed three months after mothers' participation in the study to assess whether any HPV vaccine doses were provided.

ELIGIBILITY:
Inclusion Criteria:

* Mother is greater than or equal to 18 years of age
* Mother has a daughter who is between the ages of 11-15 years
* Daughter has not received any doses of the HPV vaccine
* When asked to describe how she feels about getting her daughter vaccinated against HPV in the next six months, mother responds "I don't want her to get vaccinated" or "I'm unsure if I want her vaccinated."

Exclusion Criteria:

* Cannot read/speak English

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2010-06; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Dempsey, MD, PhD, MPH, Principal Investigator — Child Health Evaluation and Research Unit
Locations (1):
- UMHS Outpatient Pediatrics, Ann Arbor, Michigan, United States

REFERENCES:
- [Background] Centers for Disease Control and Prevention (CDC). National, state, and local area vaccination coverage among adolescents aged 13-17 years--United States, 2008. MMWR Morb Mortal Wkly Rep. 2009 Sep 18;58(36):997-1001. PMID 19763075
- [Background] Chesson HW, Blandford JM, Gift TL, Tao G, Irwin KL. The estimated direct medical cost of sexually transmitted diseases among American youth, 2000. Perspect Sex Reprod Health. 2004 Jan-Feb;36(1):11-9. doi: 10.1363/psrh.36.11.04. PMID 14982672
- [Background] Dempsey AF, Abraham LM, Dalton V, Ruffin M. Understanding the reasons why mothers do or do not have their adolescent daughters vaccinated against human papillomavirus. Ann Epidemiol. 2009 Aug;19(8):531-8. doi: 10.1016/j.annepidem.2009.03.011. Epub 2009 Apr 25. PMID 19394865
- [Background] Dempsey A, Cohn L, Dalton V, Ruffin M. Patient and clinic factors associated with adolescent human papillomavirus vaccine utilization within a university-based health system. Vaccine. 2010 Jan 22;28(4):989-95. doi: 10.1016/j.vaccine.2009.10.133. Epub 2009 Nov 17. PMID 19925899
- [Background] Dempsey AF, Zimet GD, Davis RL, Koutsky L. Factors that are associated with parental acceptance of human papillomavirus vaccines: a randomized intervention study of written information about HPV. Pediatrics. 2006 May;117(5):1486-93. doi: 10.1542/peds.2005-1381. PMID 16651301
- [Background] Gust D, Brown C, Sheedy K, Hibbs B, Weaver D, Nowak G. Immunization attitudes and beliefs among parents: beyond a dichotomous perspective. Am J Health Behav. 2005 Jan-Feb;29(1):81-92. doi: 10.5993/ajhb.29.1.7. PMID 15604052
- [Background] Hawkins RP, Kreuter M, Resnicow K, Fishbein M, Dijkstra A. Understanding tailoring in communicating about health. Health Educ Res. 2008 Jun;23(3):454-66. doi: 10.1093/her/cyn004. Epub 2008 Mar 17. PMID 18349033
- [Background] Markowitz LE, Dunne EF, Saraiya M, Lawson HW, Chesson H, Unger ER; Centers for Disease Control and Prevention (CDC); Advisory Committee on Immunization Practices (ACIP). Quadrivalent Human Papillomavirus Vaccine: Recommendations of the Advisory Committee on Immunization Practices (ACIP). MMWR Recomm Rep. 2007 Mar 23;56(RR-2):1-24. PMID 17380109

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tailoring | Untailored Information
Started | 36 | 34
Completed | 36 | 34
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tailoring | Untailored Information | Total
Number analyzed (Participants) | 36 | 34 | 70
Age, Continuous [Mean (Full Range); unit: years] | 40 [38 to 55] | 40 [32 to 60] | 40 [32 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 34 | 70
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 9 | 18
  White | 25 | 22 | 47
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 36 | 34 | 70

OUTCOME MEASURES:

1. Primary Outcome: Mother's Intention to Vaccinate Daughter Against HPV
Description: Mother will rate her intention to have her daughter vaccinated against HPV using a Likert scale before and after the intervention. The scale ranges from 0-11 with higher numbers representing more positive intentions to vaccinate against HPV, and 5 being neutral intentions (i.e. neither positive nor negative). In this assessment we use this 11-point scale to assess vaccination before and after viewing the educational materials. The difference pre and post intervention in vaccination intention is calculated (min 0, max 11) and the mean of these differences are calculated for the control and intervention groups.
Time Frame: Date of intervention (one day)
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Tailoring | Untailored Information
Number analyzed (Participants) | 36 | 34
units on a scale | 1.53 [1.31 to 1.83] | 1.29 [1.09 to 1.79]

2. Secondary Outcome: Vaccination of Daughter
Description: With mother's consent, daughter's University of Michigan vaccination record will be accessed to determine whether daughter has received any doses of the HPV vaccine. If the University of Michigan vaccination record does not document a visit three months after the intervention, with mother's consent, research staff will call mother at home to determine whether daughter has received any doses of the HPV vaccine.
Time Frame: Less than or equal to three months from the date of the intervention
Measure: Number; unit: participants
Arm/Group | Tailoring | Untailored Information
Number analyzed (Participants) | 36 | 34
participants | 1 | 2

ADVERSE EVENTS:
Time Frame: 1 day
Description: Data collected only at the time of intervention
Arm/Group | Tailoring | Untailored Information
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/34
Other Adverse Events (participants affected / at risk) | 0/36 | 0/34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes